CLINICAL TRIAL: NCT04060355
Title: Developing a Distance Education System to Train Savvy Caregiver Program Interventionists: Extending Access and Capacity in Community-Based Delivery of Evidence-Based Interventions
Brief Title: Savvy System Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kenneth Hepburn, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00108423; R01AG061971 (NIH)
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Caregiver Burnout; Dementia
Keywords: People Living With Disability; PLWD; Caregiver; Interventionist; Distance education; Savvy
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Savvy Participants (Experimental): Using an on-line survey method, each caregiver will be asked to complete the post-program fidelity monitoring survey that seeks responses to the program (feel more knowledgeable, more competent, better equipped, etc.) and asks them to assess the interventionist's performance and verify that certain key elements of the program were covered.
  Interventions: Behavioral: Savvy program
- Interventionists (Experimental): Three recorded semi-structured video interviews will be conducted with each interventionist. One will occur immediately after training; this will focus on their sense of the completeness and adequacy of the training program, including the training methods, videos, and materials, and their perceived readiness to lead the program. Another interview will be done immediately after the conduct of each of the two Savvy programs they lead, asking them to report on their performance as interventionists, including any adaptation processes in which they might have engaged, and to reflect on ways the training might be improved to strengthen their skills, including for adaptation.
  Interventions: Behavioral: Semi-structured video interviews
- Organizational Leaders (Experimental): Recorded semi-structured video interviews with sponsoring organizations' key contact persons will be conducted immediately after the interventionist training and then after each of the two Savvy offerings. The conversation will focus on identifying ways to strengthen and improve the training, certification, and fidelity monitoring system. Information about time and resource costs of the program, caregiver demand, and caregiver recruitment and feedback will be also collected.
  Interventions: Behavioral: Semi-structured video interviews

INTERVENTIONS:
Behavioral: Savvy program — Caregiver program (Savvy) is an evidence-based dementia family caregiver psychoeducation program. Provided to groups of 8-12 (typically) individuals caring for family members living with Alzheimer's disease or related dementias (PLWD), Savvy employs a mechanism of action based in Social Cognitive theory to promote caregivers' solution-focused coping behaviors through the acquisition of appropriate knowledge, skills, and outlook and the enhancement of caregiving mastery.
  Arms: Savvy Participants
Behavioral: Semi-structured video interviews — Semi-structured video interviews will assess the preliminary efficacy of programs led by system-trained interventionists in producing anticipated outcomes in caregiver participants - reduced depression and burden and enhanced caregiving mastery. It will also focus on sense of the completeness and adequacy of the training program, including the training methods, videos, and materials
  Arms: Interventionists; Organizational Leaders

SUMMARY:
The study goal is to develop a web-based system that uses distance education methods and provides manuals and protocols to train, certify, and monitor the performance of interventionists to deliver the Savvy Caregiver program (Savvy), an evidence-based dementia family caregiver psychoeducation program. The system has a potential to increase the scalability of Savvy.

DETAILED DESCRIPTION:
The number of People Living With Disability (PLWD) in the U.S. will rise from 5.7 million to 14 million by 2050, and the number of family caregivers who maintain these persons in the community will rise proportionately from 15 million at present. Several psychoeducation programs, including Savvy, have successfully ameliorated the adverse effects of caregiving, but these programs are only minimally available and accessible.

The study goal is to develop a web-based system that uses distance education methods and provides manuals and protocols to train, certify, and monitor the performance of interventionists to deliver the Savvy Caregiver program (Savvy), an evidence-based dementia family caregiver psychoeducation program. The system has a potential to increase the scalability of Savvy.

ELIGIBILITY:
Inclusion Criteria:

Organizational Leaders

1. Able to understand and speak English
2. Affiliated with an organization serving caregivers for family members living with Alzheimer's disease or related dementias
3. 18 years or older

Interventionists

1. Able to understand and speak English
2. Affiliated with a participating organization
3. 18 years or older

Caregivers

1. Able to understand and speak English
2. Caregiver for a person living with Alzheimer's disease or related dementias (PLWD) who is providing informal care for at least 3 hours a day. PLWD should not be bound for institutional care within the next 6 months.
3. 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hepburn, PhD, Principal Investigator — Emory University
Locations (1):
- School of Nursing, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication, up to 5 years after publication
Access Criteria: Researchers who provide a methodologically sound proposal should submit request to khepbur@emory.edu. Requesters will be required to complete and sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 family caregivers who took part in Savvy Caregiver programs led by interventionists trained by the online training program developed in this project consented to be part of the study and provided baseline data. These caregivers were recruited from 37 Savvy Caregiver programs offered by 23 of the trained interventionists from 13 agencies located in 5 states. The first caregiver enrolled on 8/04/21. The last caregiver data collection point occurred on 09/27/2023
Period: Overall Study
Arm/Group | Savvy Participants
Started | 120
Completed | 79 (41 of those who provided baseline data did not, despite repeated attempts to reach them, reply to requests to schedule the 6-month interviews)
Not Completed | 41
Not completed — Lost to Follow-up | 41

BASELINE CHARACTERISTICS:
Arm/Group | Savvy Participants
Number analyzed (Participants) | 120
Age, Customized [Mean (Standard Deviation); unit: years]
  Age 33- 83 | 67.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 111
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 105
  More than one race | 0
  Unknown or Not Reported | 6
Relationship to PLWD (People living with Dementia) [Count of Participants; unit: Participants]
  Spouse | 70
  Child/ Other Relative | 43
  Sibling/ Friend/ Other | 7
Live with PLWD: Yes [Count of Participants; unit: Participants] | 91
Employed outside home: No [Count of Participants; unit: Participants] | 88
Any other help with caregiving: Yes [Count of Participants; unit: Participants] | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in Center for Epidemiologic Studies - Depression Scale (CES-D) Score
Description: The CES-D scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past week. It includes 20 items comprising six scales reflecting major facets of depression: depressed mood, feelings of guilt and worthlessness, feelings of helplessness and hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Savvy Participants
Number analyzed (Participants) | 120
score on a scale
  Baseline | 13.2 (9.1)
  Month 6 | 79 (11.0)

2. Secondary Outcome: Change in Anxiety Score
Description: State-Trait Anxiety Inventory scale - 20-item 4-point Likert scale is sensitive to changes in transitory anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" (0) to "Almost Always" (3)); Range: 0-60. Higher scores indicate greater anxiety.
Time Frame: Baseline, Month 6
Population: The analysis population includes participants who completed the required assessment at follow-up appointments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Savvy Participants
Number analyzed (Participants) | 120
score on a scale
  Baseline | 34.9 (10.2)
  Month 6 | 35.3 (11.5)

3. Secondary Outcome: Change in Zarit Burden Inventory (ZBI) Score
Description: Zarit Burden Inventory (ZBI) score is a 22-item Likert scale. Each item is a statement which the caregiver is asked to endorse using a 5-point scale, scored "Never" (0) to "Nearly Always" (4); Range: 0-88. Total score is obtained by summing all items endorsed. Higher scores indicate greater perceived burden.
Time Frame: Baseline, Month 6
Population: The analysis population includes participants who completed the required assessment at follow-up appointments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Savvy Participants
Number analyzed (Participants) | 120
score on a scale
  Baseline | 35.9 (14.2)
  Month 6 | 35.2 (13.4)

4. Secondary Outcome: Change in Caregiver Pearlin Mastery Score
Description: The Pearlin Mastery (PM) scale measures the extent to which an individual regards their life chances as being under their personal control rather than fatalistically ruled. Response options: 4-point Likert scale, 1,"Strongly disagree" and 4,"Strongly agree". Items are summed, yielding a range from 7 to 28. Higher scores indicate greater levels of mastery.
Time Frame: Baseline, Month 6
Population: The analysis population includes participants who completed the required assessment at follow-up appointments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Savvy Participants
Number analyzed (Participants) | 120
score on a scale
  Baseline | 11.5 (2.1)
  Month 6 | 12.7 (1.6)

5. Secondary Outcome: Change in Revised Memory and Behavior Problem Checklist Score
Description: Revised Memory and Behavior Problem Checklist is a 24-item two-part Likert scale that assesses (Part 1) caregiver reported frequency of patient behaviors and (Part 2) caregiver's responreaction to each behavior, or the extent of distress experienced. The frequency of behaviors is assessed based on a Likert-scale of 0 to (0 = never occurs, 1 = occurs infrequently and not in the last week, 2 = occurred 1-2 times in the last week, 3 = occurred 3-6 times in the last week, and 4 = occurs daily or more often); Range: 0-96. Reactions are assessed by asking how" upsetting" the behavior was on a Likert scale of 0 to 4 (0 = Not at all, 1= a little, 2 = moderately, 3 = very much, and 4 =extremely); Range: 0-96. The two parts of the scale yield a summary score - higher scores indicate higher frequency of patient behaviors and greater levels of caregiver distress, respectively.
Time Frame: Baseline, 6 months
Population: The analysis population includes participants who completed the required assessment at follow-up appointments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Savvy Participants
Number analyzed (Participants) | 120
score on a scale
  Baseline Frequency | 38.7 (12.2)
  Month 6 Frequency: number analyzed (Participants) | 78
  Month 6 Frequency | 36.6 (11.8)
  Baseline Reaction | 19.7 (11.9)
  Month 6 Reaction: number analyzed (Participants) | 78
  Month 6 Reaction | 17.0 (11.0)

ADVERSE EVENTS:
Time Frame: : Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Month 12
Arm/Group | Savvy Participants
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

LIMITATIONS AND CAVEATS:
The study was not conducted as a two-armed trial as originally planned; therefore, there is no second group for data reporting. Most of the project occurred during the COVID pandemic, especially the caregiver component. Collaborating agencies were unwilling to suggest that clients volunteer for a trial requiring a 4-month wait for the Savvy Caregiver program. Due to recruitment challenges, the trial was run as a one-arm, collecting data at baseline and 6 months instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT04060355/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04060355/ICF_000.pdf